CLINICAL TRIAL: NCT05691270
Title: IN Control: Contraception Navigator Program for Adolescents and Young Adults in Indiana
Brief Title: Contraception Navigator Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Tracey Wilkinson, Assistant Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1801682245; 5K23HD094853-04 (NIH)
Record Dates: First submitted 2022-11-23; First posted 2023-01-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Contraception; Contraceptive Usage; Health Care Utilization
Keywords: Birth Control Access; Access; Navigator
MeSH Terms: conditions — Contraception Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: All adolescents who engage with the IN-Control program will be asked if they would like to formally enroll as a study participant after interaction with the navigator; however, enrollment is not required to utilize the services of the navigator,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Study Participants (Other): All adolescents who engage with the IN-Control Program will be asked if they would like to formally enroll as a study participant after interaction with the navigator. However, enrollment is not required to receive support from the navigator.
  Interventions: Behavioral: IN-Control (Birth Control Navigator Program)

INTERVENTIONS:
Behavioral: IN-Control (Birth Control Navigator Program) — Pilot Study of IN-Control Program within the state of Indiana

SUMMARY:
The goal of this study is to pilot test the IN-Control Birth Control Navigator Program in Central Indiana for use by adolescents who would like to access birth control. The investigators hypothesize that facilitating access to contraception through our intervention will ultimately result in increased feelings of autonomy around these decisions and use of hormonal contraception.

DETAILED DESCRIPTION:
The IN-Control Birth Control Navigator Program will provide personalized attention to adolescents and young adults and will be able to address self-efficacy skills, and abilities through personal interactions with navigator staff and use of targeted services. Importantly, the navigator can assist participants in overcoming specific environmental barriers (transportation, cost, clinical access) and personal barriers (knowledge and confidentiality concerns) before, during and after the clinical encounter.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 15-19 yrs
* English speaking
* Lives in Indiana

Exclusion Criteria:

* Adolescents younger than 15 or older than 19 yrs
* Non-English speaking
* Lives outside of Indiana

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — We anticipate females accessing our program that are in need of hormonal birth control.
Enrollment: 35 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction with IN Control Program (feeling comfortable, listened to, helpful, easy to contact) | Within 2-4weeks after contact with the IN-Control Program
  Survey of participants that interacted with navigator program (percentage of participants reporting that the navigator program was easy to contact, made them feel comfortable, listened to and helpful)

SECONDARY OUTCOMES:
Navigator Inquiries | Duration of Pilot Study, 2 years
  Number of unique individuals contacting navigator program
Website Utilization | Duration of Pilot Study, 2 years
  Number of unique website visits
Birth Control Decision Aid | Duration of Pilot Study, 2 years
  Completion Rate of My Birth Control Decision Aid
Contact Success Rate | Duration of Pilot Study, 2 years
  number of individuals endorsing wanting additional help from navigator staff compared to the number of individuals successfully contacted by navigator staff

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is no current plan to share the data with any other researchers.

REFERENCES:
- [Background] Wilkinson TA, Hawryluk B, Moore C, Peipert JF, Carroll AE, Wiehe S, Fortenberry JD. Developing a Youth Contraception Navigator Program: A Human-Centered Design Approach. J Adolesc Health. 2022 Aug;71(2):217-225. doi: 10.1016/j.jadohealth.2022.03.005. Epub 2022 May 11. PMID 35562301
- [Background] Wilkinson TA, Hawryluk B, Moore C, Peipert JF, Carroll AE, Wiehe S, Fortenberry JD. A human-centered designed outreach strategy for a youth contraception navigator program. PEC Innov. 2022 Dec;1:100093. doi: 10.1016/j.pecinn.2022.100093. Epub 2022 Oct 18. PMID 36540664
- See also: Program Website — http://www.in-control.me